CLINICAL TRIAL: NCT01672749
Title: Evaluation of a Growth Guiding Construct vs. Standard Dual Growing Rods and VEPTR for the Treatment of Early Onset Scoliosis Patients: A Prospective Multi-center Cohort Study With a Matched Historical Control
Brief Title: Evaluation of a Modern System to Allow for Growth in Children With Scoliosis Versus a Conventional Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: EOS TROLLEY
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Early Onset Scoliosis
Keywords: Scoliosis [MESH]; Pediatrics [MESH]; Early onset; Growth guidance; Growing rod; Trolley; Dual growing rod technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Spine based dual growing rod or VEPTR: Patients treated with the TROLLEY system will be compared with patients from the Chest Wall and Spine Deformity Study Group (CWSDSG) and the Growing Spine Study Group (GSSG) treated with a spine based dual growing rod or the rib based Vertical Expandable Prosthetic Titanium Rib (VEPTR, Synthes North America). For each patient in the TROLLEY group a patient from each of the databases will be selected to be matched based on diagnosis, age, gender, and spine deformity classification.
  Interventions: Device: Spine based dual growing rod or rib based VEPTR
- TROLLEY system: Growth guiding construct using the DePuy Synthes TROLLEY Gliding Vehicles (GVs). The TROLLEY system is CE marked at the time of the study conduct.
  Interventions: Device: Growth guiding construct using TROLLEY system

INTERVENTIONS:
Device: Growth guiding construct using TROLLEY system — Growth guiding construct using the DePuy Synthes TROLLEY Gliding Vehicles (GVs)
  Groups: TROLLEY system
Device: Spine based dual growing rod or rib based VEPTR — spine based dual growing rod or the rib based Vertical Expandable Prosthetic Titanium Rib (VEPTR, Synthes North America)
  Groups: Spine based dual growing rod or VEPTR

SUMMARY:
The foremost challenge when managing early onset scoliosis (curve deformity before the age of 10) is to prevent curve progression while maintaining growth of the spine. Current treatment options require repetitive interventions as the spine and the child grow. This study will compare two techniques of growth modulation: Standard dual growing rods versus the new Luqué Trolley screws

Hypothesis: Patients treated with the DePuy Synthes TROLLEY system will undergo fewer re-operations after 3 years of follow-up (FU) than patients included in the comparison group

DETAILED DESCRIPTION:
The purpose of this clinical study is to show that the growth guiding construct with DePuy Synthes TROLLEY Gliding Vehicles allows for less re-operations and for ongoing spinal growth across an instrumented immature spine while preventing curve progression in early onset scoliosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 - 10 years
* Diagnosis of Early Onset Scoliosis with any of the following etiologies:

Idiopathic Congenital Neuromuscular Syndromic Mesenchymal

- Significant growth potential defined by any of the following: pre peek growth velocity bone age < 10; open triradiate cartilage

* An expected significant spinal deformity of more than 80 degrees at skeletal maturity
* Signed informed consent as legally required (patient, parents, etc.)
* Willingness and ability of the patient to participate in the clinical investigation including imaging and FU procedures
* Willingness and ability of the parents to support the patient in his/her study participation
* Ability of the patient and parents to understand the content of the patient information / informed consent form and participate in the clinical investigation
* Signed informed consent by patient / parent(s)

Exclusion Criteria:

* Curve magnitude and rigidity: Cobb greater than 100 degrees or bends less than 50 degrees
* Prior spinal surgery
* Skeletal maturity
* Any not medically managed severe systemic disease
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: One third of the patients will be recruited in designated investigation sites using the TROLLEY system. For each trolley patient one to two comparative matched pairs will be generated from mining the database of the Chest Wall and Spine Deformity Study Group (CWSDSG) and the Growing Spine Study Group (GSSG).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2023-02 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Number of re-operations | 3 years FU
  Number of re-operations of the spine per patient in both groups after 3 years of FU

SECONDARY OUTCOMES:
Sitting height | 10 years
Standing height | 10 years
Radiographic measurements | 10 years
  * Spine length: upper T1 to lower L5 end plates
  * Chest length: upper T1 to Lower T12
  * Instrumented spine length
Curve / deformity type characteristics | 10 years
  * Lenke classification
  * New EOS classification
Adverse Events related to the procedure and/or device under investigation | 10 years
Quality of life | 10 years
  * EOS Questionnaire (EOSQ 24)
  * Pediatric version of EQ-5D (EQ-5D-Y)
Pulmonary function: | 10 years
  * Forced vital capacity (FVC), actual [L] and predicted [%]
  * Forced expiratory volume in 1 second (FEV1), actual [L] and predicted [%]
  * Total lung capacity (TLC), actual [L] and predicted [%]
  * Use and rate of assisted ventilation
  * Residual volume (RV)
Growth potential | 10 years
  * Chronological age
  * Bone age (based on radiograph of the hand)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Ouellet, MD, Principal Investigator — McGill University Health Science Centre, Montreal, Canada
Locations (3):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland
- United Kingdom (2):
  - Queen's Medical Centre, Nottingham
  - Sheffield Children's Hospital, Sheffield

REFERENCES:
- [Derived] Dayer R, Grevitt M, Breakwell L, Yoon W, Chen M, Ratz T, Szocik T, Zhu YY; Pediatric Spine Study Group (PSSG); Ouellet J. Management of early-onset scoliosis: modern Luque trolley technique led to fewer reoperations within 3 years than other growth-friendly techniques, a prospective cohort study with matched historical controls. Spine Deform. 2025 Sep;13(5):1611-1624. doi: 10.1007/s43390-025-01102-2. Epub 2025 May 28. PMID 40437325